CLINICAL TRIAL: NCT01150513
Title: Docetaxel Plus Carboplatin Versus Epirubicin Plus Cyclophosphamide Followed by Docetaxel as Adjuvant Treatment in Triple-negative Breast Cancer
Brief Title: Docetaxel+Carboplatin vs Epirubicin+Cyclophosphamide Followed by Docetaxel as Adjuvant Treatment in Triple-negative Breast Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-007
Record Dates: First submitted 2010-06-14; First posted 2010-06-25 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: TRIPLE-NEGATIVE; BREAST CANCER
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EC-T (Active Comparator)
  Interventions: Drug: EC-T
- TP (Experimental)
  Interventions: Drug: TP

INTERVENTIONS:
Drug: EC-T — four cycles of EC (epirubicin: 90 mg/m2; cyclophosphamide :600 mg/m2, day 1) followed by four cycles of T (docetaxel : 75 mg/m2 or paclitaxel 175 mg/m2, day 1)
  Arms: EC-T
Drug: TP — six cycles of TP (docetaxel: 75 mg/m2 or paclitaxel 175 mg/m2 d1; carboplatin AUC=5, day 1)
  Arms: TP

SUMMARY:
Triple-negative breast cancer (TNBC) has a relatively bad prognosis whereas there is no standard regimen. Some data showed that platins could improve the efficacy of advance TNBC. In this trial, it is the hypothesis that TP (docetaxel plus carboplatin) has a better efficacy than EC-T (epirubicin plus cyclophosphamide followed by docetaxel).

ELIGIBILITY:
Inclusion Criteria:

* Triple-negative breast cancer
* Older than 18 years old
* Have tumor resection surgery
* Sufficient organ function (marrow, heart, liver)

Exclusion Criteria:

* Other malignancy
* Other serious disease( marrow, heart, liver)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2009-06; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) of 3 years | 3 years after mastectomy
  local recurrence, distant metastasis, the secondary primary malignancy

SECONDARY OUTCOMES:
Safety Profiles | Up to 24 weeks
  All adverse events occurring during chemotherapy are to be recorded in the case report form, including hemotologic and nonhemotologic toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Chen Y, Wang X, Du F, Yue J, Si Y, Zhao X, Cui L, Zhang B, Bei T, Xu B, Yuan P. Association between homologous recombination deficiency and outcomes with platinum and platinum-free chemotherapy in patients with triple-negative breast cancer. Cancer Biol Med. 2023 Mar 2;20(2):155-68. doi: 10.20892/j.issn.2095-3941.2022.0525. PMID 36861447
- [Derived] Zheng F, Du F, Wang W, Wang Y, Li M, Zhao J, Wang X, Yue J, Wang J, Yang Z, Cai R, Ma F, Fan Y, Li Q, Zhang P, Xu B, Yuan P. Updated efficacy of adjuvant epirubicin plus cyclophosphamide followed by taxanes versus carboplatin plus taxanes in early triple-negative breast cancer in phase 2 trial: 8.1-year median follow-up. Breast Cancer Res Treat. 2022 Jan;191(1):97-105. doi: 10.1007/s10549-021-06401-6. Epub 2021 Oct 14. PMID 34648118